CLINICAL TRIAL: NCT06869811
Title: Oral Anticoagulation Versus Left Atrial Appendage Occlusion Added to Direct Oral Anticoagulation in Patients with Stroke Despite Oral (ADD-LAAO TRIAL)
Brief Title: Oral Anticoagulation Versus Left Atrial Appendage Occlusion Added to Direct Oral Anticoagulation in Patients with Stroke Despite Oral
Acronym: ADDLAAO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital San Carlos, Madrid (Other); Hospital Álvaro Cunqueiro (Other); Hospital Universitari de Bellvitge (Other); University of Salamanca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADD-LAAO
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-07

CONDITIONS: Left Atrial Appendage Closure
Keywords: LAAO; Stroke; Oral Anticoagulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: 2 arms
  Treatment vs. Procedure + treatment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Best medical treatment (Active Comparator): The best medical treatment selected by the neurologist including change OAC/DOAC or intensification of the antithrombotic treatment.
  Interventions: Device: LAA Closurse
- Left atrial appendage occlusion + DOAC or OAC (Active Comparator): LAA Occlusion + DOAC (unless there is a compelling use of OAC like in a mechanical valve).
  Interventions: Device: LAA Closurse

INTERVENTIONS:
Device: LAA Closurse — LAA Closure + DOAC or OAC

SUMMARY:
A total of 380 patients with ischemic stroke despite OAC will be included. Patients will be randomized 1:1 to the best medical treatment (control) or the combination of LAAO and DOAC or OAC. The study's primary endpoint will be the occurrence of a cardioembolic event (ischemic stroke or arterial peripheral embolism) within the first 12 months after inclusion.

DETAILED DESCRIPTION:
Background: The prevalence of atrial fibrillation and the number of patients experiencing ischemic strokes despite being on oral anticoagulation (OAC) are both increasing. This rise presents a significant challenge due to the absence of clear and uniform treatment recommendations for these patients. To date, there is no formal combination that merges a high anticoagulant efficacy while keeping a low bleeding risk. Transcatheter left atrial appendage occlusion (LAAO) added to OAC might provide a balance between efficacy and safety.

Objectives: To evaluate if, in patients with ischemic stroke despite OAC, the combination of LAAO and long-term direct OAC (DOAC) or OAC is associated with a lower incidence of recurrent cardioembolic events at 12 months as compared to the best medical treatment proposed by the neurologist.

Methods: A total of 380 patients with ischemic stroke despite OAC will be included. Patients will be randomized 1:1 to the best medical treatment (control) or the combination of LAAO and DOAC or OAC. The study's primary endpoint will be the occurrence of a cardioembolic event (ischemic stroke or arterial peripheral embolism) within the first 12 months after inclusion.

Implication: This study is one of the first randomized trials comparing the LAAO+DOAC combination to optimal medical treatment in patients who have had ischemic strokes despite being on OAC. If the results confirm the superiority of LAAO+DOAC, it could lead to a paradigm shift in treatment guidelines for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Cardioembolic* Ischemic stroke despite OAC or DOAC within the last 6 months.
* Documented AF (either valvular or non-valvular AF).
* LAA suitable for closure (if LAA thrombus, just distal).
* Functional status at inclusion with no severe disability (mRS<4).
* No contraindication for LAA assessment by CT or 3D-TEE.
* >18 years
* Life expectancy >1year
* Able to understand written consent prior to the trial inclusion.
* Able and willing to return for follow-up visits and tests.

Exclusion Criteria:

* Absolute contraindication to OAC/DOAC.
* Non-compliance of OAC/DOAC >24 hours within the last week before the index stroke (>1 dose per - - Antagonist Vit K and >2 doses per DOAC).
* Lacunar Ischemic Stroke.
* Symptomatic carotid disease (defined as > 50% lumen diameter narrowing on CTA, MRA, or TCD with symptoms of ipsilateral transient or visual TIA evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke); if subject has a history of carotid stent or endarterectomy the subject is eligible if there is < 50% lumen diameter narrowing.
* Planned cardiac intervention or surgery, which is invasive or requires sedation or anesthesia, within 3 months following randomization, other than study-related procedures such as LAAO and cardiac imaging (if applicable).
* In the opinion of the investigator, is considered at high risk for general anesthesia and general anesthesia is planned for the study procedure.
* Non-treated patent foramen ovale (PFO) or PFO closure device implanted.
* Inferior vena cava filter.
* Has any of the customary contraindications for a percutaneous catheterization procedure (e.g. subject is too small to accommodate the ICE probe (if planned) or required catheters, or subject has - active infection or bleeding disorder).
* Customary contraindications for TEE/TOE (e.g., presence of esophageal varices, esophageal stricture, or history of esophageal cancer).
* Underwent catheter ablation for AF or atrial flutter within 60 days prior to randomization.
* Experienced myocardial infarction within 90 days prior to randomization.
* New York Heart Association Class IV Congestive Heart Failure.
* Left ventricular ejection fraction ≤ 30% (per most recent assessment).
* LAA is obliterated or surgically ligated.
* Thrombocytopenia (defined as < 50,000 platelets per microliter (<50 x 109/L) or anemia (defined as hemoglobin < 10 g/dL) requiring transfusions.
* Hypersensitivity to any portion of the device material or individual components of the Amulet LAA occluder device (e.g., nickel allergy).
* Allergy to contrast media if the patient needs angio-CT and cannot undergo TEE/TOE.
* Actively enrolled in, or plans to enroll in, a concurrent clinical study in which the active treatment arm may confound the results of this trial.
* Is pregnant or breastfeeding, or pregnancy is planned during the course of the investigation.
* Active endocarditis or other infection producing bacteremia.
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the Investigator's opinion, could limit the subject's ability to participate in clinical investigation or to comply with follow up requirements, or impact the scientific soundness of the clinical investigation results.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-07-22 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 12 months
  The study's primary endpoint will be the occurrence of a cardioembolic event (ischemic stroke or arterial peripheral embolism) within the first 12 months after inclusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided